CLINICAL TRIAL: NCT02806726
Title: A Prospective Study to Evaluate the Feasibility of a New Treatment Algorithm to Increase Depth of Focus After Wavefront-guided LASIK Correction of Myopic Refractive Errors With the iDesign System and Star S4 IR™ Excimer Laser System
Brief Title: Clinical Investigation iDesign System With 1.3-PRESBY Treatment and STAR S4 IR™ Excimer Laser System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision to discontinue product development at this time
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAR-116-TOPS
Record Dates: First submitted 2016-06-08; First posted 2016-06-21 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Presbyopia; Myopia
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- iDesign 1.3-PRESBY (Experimental): iDesign 1.3-PRESBY in one eye of subject (experimental) is used to calculate the LASIK treatment profile for the iDesign Advanced Wavescan Studio™ System within the Star S4 IR™ Excimer Laser System.
  Interventions: Device: iDesign 1.3-PRESBY treatment
- iDesign 1.3 (Active Comparator): iDesign 1.3 in one eye of subject (control) is used to calculate the LASIK treatment profile for the iDesign Advanced Wavescan Studio™ System within the Star S4 IR™ Excimer Laser System.
  Interventions: Device: iDesign 1.3 treatment

INTERVENTIONS:
Device: iDesign 1.3-PRESBY treatment — Software used to calculate the LASIK treatment profile including a presbyopic correction component for the iDesign Advanced Wavescan Studio™ System within the Star S4 IR™ Excimer Laser System.
  Arms: iDesign 1.3-PRESBY
Device: iDesign 1.3 treatment — Software used to calculate the LASIK treatment profile for the iDesign Advanced Wavescan Studio™ System within the Star S4 IR™ Excimer Laser System.
  Arms: iDesign 1.3

SUMMARY:
A prospective study to evaluate the feasibility of a new treatment algorithm to increase depth of focus after wavefront-guided LASIK correction of myopic refractive errors with the iDesign Advanced Wavescan Studio™ System and Star S4 IR™ Excimer Laser System. The purpose of this study is to determine whether wavefront-guided LASIK correction of myopic refractive errors with CustomVue combined with iDesign 1.3-PRESBY (presbyT-LASIK) treatments mitigate the effects of presbyopia by increasing the depth of focus compared to iDesign CustomVue treatments.

ELIGIBILITY:
Inclusion Criteria:

All criteria apply to each eye

1. Signed informed consent and Personal Health Information Protection Act authorization.
2. At least 45 years of age at enrollment (date informed consent signed).
3. The refractive error, based on the iDesign displayed refraction selected for treatment ("4.0 Rx calc" at 12.5 mm), must be myopia with or without astigmatism with sphere up to -6.00 D, and cylinder between 0.00 D and -5.00 D with a maximum spherical equivalent (SE) of -8.00 D.
4. Require an add power of +1.00 D or more during near testing at 40 cm.
5. Anticipated stromal bed thickness of at least 250 microns based on preoperative central corneal pachymetry minus the maximum ablation depth (as calculated by the iDesign system) plus the intended flap thickness.
6. Distance Best Spectacle Corrected Visual Acuity (BSCVA) of 20/20 or better.
7. Uncorrected Visual Acuity (UCVA) of 20/40 or worse.
8. Less than or equal to 0.75 D difference between cycloplegic and manifest refraction sphere.
9. A stable refractive error (based on a previous exam, medical records, lensometry, or prescription at least 12 months prior to the preoperative manifest refraction), as defined by a change of ≤1.00 D in MRSE.
10. Any eye with a history of contact lens wear within the last 4 weeks must demonstrate refractive stability according to the following:

    1. Rigid contact lenses (toric or spherical) must be removed for at least 4 weeks and soft contact lenses (toric or spherical) for at least 2 weeks prior to the first refraction used to establish stability.
    2. Two consecutive refractions and keratometric readings must be conducted at least 7 days apart.
    3. Refractive stability is defined as a change of not more than 0.50 D in manifest refraction sphere and cylinder as well as mean keratometry between measurements.
    4. If the subject/eye meets the refractive stability criteria, contact lens wear is not permitted prior to surgery.
11. Agreement between manifest refraction (adjusted for optical infinity) and iDesign System refraction chosen for treatment, as follows:

    1. Spherical Equivalent: Magnitude of the difference is less than 0.625 D.
    2. Cylinder: Magnitude of the difference is less than or equal to 0.5 D.
    3. Cylinder Axis Tolerance: If either the manifest cylinder entered into the iDesign System or the iDesign cylinder selected for treatment is less than 0.5 D, there is no requirement for axis tolerance. When both cylinders have a magnitude of at least 0.5 D, the axis tolerance as determined by the iDesign system is linearly reduced from 15 (0.5 D) to 7.5 (7.0 D) based on the average magnitude of both cylinders. Note: If the axis tolerance is not in the calculated range, the iDesign system will produce a warning and this exam may not be used for treatment planning.
12. Willing and capable of complying with follow-up examinations for the duration of the study.

Exclusion Criteria:

1. Women who are pregnant, breast-feeding, intend to become pregnant, or are not using an adequate method of birth control [examples are any form of barrier contraception (such as condom or diaphragm with contraceptive cream/jelly), birth control pills, hormonal implant, IUD, abstinence or surgical sterilization (tubal ligation, hysterectomy or vasectomy)]. Note: Women who were pregnant or nursing may not be enrolled until 6 months after either delivery or have stopped nursing and there is documented refractive stability.
2. Concurrent use of systemic (including inhaled) medications that may impair healing, including but not limited to: antimetabolites, isotretinoin (Accutane®) within 6 months of treatment, and amiodarone hydrochloride (Cordarone®) within 12 months of treatment.

   NOTE: The use of inhaled or systemic corticosteroids, whether chronic or acute, is deemed to adversely affect healing and subjects using such medications are specifically excluded from eligibility.
3. History of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or herpes simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis.

   NOTE: The presence of diabetes (either type 1 or 2), regardless of disease duration, severity, or control, will specifically exclude subjects from eligibility.
4. Subjects with a cardiac pacemaker, implanted defibrillator or other implanted electronic device.
5. History of prior intraocular or corneal surgery (including cataract extraction), active ophthalmic disease or abnormality (including, but not limited to, symptomatic blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1 mm from limbus), retinal detachment/repair, clinically significant lens opacity, clinical evidence of trauma, corneal opacity within the central 9 mm and visible on topography, at risk for developing strabismus, or with evidence of glaucoma or propensity for narrow angle glaucoma.

   NOTE: Subjects with open angle glaucoma, regardless of medication regimen or control, or an IOP greater than 21 mmHg at screening, are specifically excluded from eligibility.
6. Evidence of keratoconus, corneal dystrophy or irregularity, or abnormal topography.
7. Known sensitivity or inappropriate responsiveness to any of the medications used in the postoperative course.
8. Desire to have monovision.
9. Intolerance to multifocal correction based on questionnaire responses to contact lens trial.
10. Participation in any other clinical study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Hileman, Study Director — Abbott Medical Optics

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per the protocol, the total number of participants enrolled is 42 (the number of participants who agreed to participate in the study and completed the informed consent process). The total number of participants Started is 7 (the number of participants who were assigned to each Arm/Group).
Units Other Than Participants: Eyes Treated
Groups:
- All Study Participants: Parts of a participant were allocated to different interventions:
  1. Left side iDesign 1.3-PRESBY, Right side iDesign 1.3
  2. Left Side iDesign 1.3, Right Side iDesign 1.3-PRESBY
Period: Overall Study
Arm/Group | All Study Participants
Started | 7; 14 Eyes Treated (Subjects were treated contralaterally)
Completed | 6; 12 Eyes Treated (Subjects were treated contralaterally)
Not Completed | 1; 2 Eyes Treated
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The safety population will be the primary analysis population for all endpoints and includes all eyes that receive study treatment.
Units Other Than Participants: Eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Number analyzed (Eyes) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) at 67 cm
Description: Mean distance corrected intermediate visual acuity (DCIVA) for presbyT-LASIK treatments (test) was compared to iDesign CustomVue treatments (control).
Time Frame: 6 months
Population: Due to the small sample size, descriptive results for all endpoints are provided along with confidence intervals, and no statistical conclusions are made.
Measure: Mean (95% Confidence Interval); unit: LogMAR
Units Other Than Participants: Eyes
Groups:
- iDesign 1.3-Presby Treatment (Experimental): One of subject's eye (experimental) treated with wavefront-guided LASIK correction of myopic refractive errors with the iDesign Advanced Wavescan Studio™ System with iDesign 1.3-PRESBY (presbyT-LASIK) treatments
- iDesign CustomVue Treatments (Control): One of subject's eye (control) treated with wavefront-guided LASIK correction of myopic refractive errors with the iDesign Advanced Wavescan Studio™ System with iDesign CustomVue treatments
Arm/Group | iDesign 1.3-Presby Treatment (Experimental) | iDesign CustomVue Treatments (Control)
Number analyzed (Participants) | 6 | 6
Number analyzed (Eyes) | 6 | 6
LogMAR | 0.03 [-0.1 to 0.16] | 0.1 [-0.02 to 0.22]

2. Secondary Outcome: Monocular Distance Corrected Near Visual Acuity (DCNVA) AT 40 cm
Description: Mean distance corrected near visual acuity (DCNVA) for PresbyT-LASIK treatments (test) was compared to iDesign CustomVue treatments (control).
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: LogMar
Units Other Than Participants: Eyes
Arm/Group | iDesign 1.3-Presby Treatment (Experimental) | iDesign CustomVue Treatments (Control)
Number analyzed (Participants) | 6 | 6
Number analyzed (Eyes) | 6 | 6
LogMar | 0.25 [0.16 to 0.34] | 0.35 [0.1 to 0.6]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=7)
Diffuse lamellar keratitis (Eye disorders) | 1 — in iDesign 1.3-Presby Treated Eye
Mild Headache (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.

DOCUMENTS (2):
  • Study Protocol (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT02806726/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT02806726/SAP_001.pdf